CLINICAL TRIAL: NCT01540825
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 113608 in Healthy Male Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: First in Man Trial of BI 113608
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1314.1; 2011-005034-19 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-02-13; First posted 2012-02-29 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Healthy

ARMS (11):
- BI 113608 high dose 1 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 low dose 1 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 low dose 2 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 low dose 4 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 low dose 5 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 medium dose 1 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 medium dose 2 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 medium dose 3 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 high dose 2 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- BI 113608 high dose 3 (Experimental): Powder for oral solution
  Interventions: Drug: BI 113608
- Placebo (Placebo Comparator): Powder for oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 113608 — Low dose powder for oral solution
  Arms: BI 113608 low dose 1
Drug: BI 113608 — High dose powder for oral solution
  Arms: BI 113608 high dose 1
Drug: BI 113608 — Medium dose powder for oral solution
  Arms: BI 113608 medium dose 3
Drug: BI 113608 — Low dose powder for oral solution
  Arms: BI 113608 low dose 2
Drug: Placebo — Powder for oral solution
  Arms: Placebo
Drug: BI 113608 — Low dose powder for oral solution
  Arms: BI 113608 low dose 5
Drug: BI 113608 — High dose powder for oral solution
  Arms: BI 113608 high dose 2
Drug: BI 113608 — High dose powder for oral solution
  Arms: BI 113608 high dose 3
Drug: BI 113608 — Medium dose powder for oral solution
  Arms: BI 113608 medium dose 1
Drug: BI 113608 — Medium dose powder for oral solution
  Arms: BI 113608 medium dose 2
Drug: BI 113608 — Low dose powder for oral solution
  Arms: BI 113608 low dose 4

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 113608 in healthy male volunteers following oral administration of single rising doses.

A secondary objective is the exploration of the pharmacokinetics of BI 113608 after single dosing.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a single dose of a placebo oral solution of volume matching the respective dose group
- BI 113608 0.5mg: Participants received a single dose of BI 113608 0.5mg powder for oral solution
- BI 113608 1mg: Participants received a single dose of BI 113608 1mg powder for oral solution
- BI 113608 2mg: Participants received a single dose of BI 113608 2mg powder for oral solution
- BI 113608 5mg: Participants received a single dose of BI 113608 5mg powder for oral solution
- BI 113608 10mg: Participants received a single dose of BI 113608 10mg powder for oral solution
- BI 113608 20mg: Participants received a single dose of BI 113608 20mg powder for oral solution
- BI 113608 50mg: Participants received a single dose of BI 113608 50mg powder for oral solution
- BI 113608 100mg: Participants received a single dose of BI 113608 100mg powder for oral solution
- BI 113608 150mg: Participants received a single dose of BI 113608 150mg powder for oral solution
- BI 113608 200mg: Participants received a single dose of BI 113608 200mg powder for oral solution
Period: Overall Study
Arm/Group | Placebo | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Started | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomised subjects who received 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg | Total
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (10.0) | 29.2 (8.1) | 34.8 (6.4) | 36.8 (12.8) | 28.5 (9.5) | 41.2 (4.6) | 30.5 (9.6) | 37.2 (11.8) | 39.7 (11.7) | 35.3 (11.3) | 38.8 (9.2) | 35.9 (10.0)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 80

OUTCOME MEASURES:

1. Primary Outcome: Clinically Relevant Abnormalities for Clinical Laboratory Evaluation, Vital Signs, Lung Function, Carbon Monoxide Diffusing Capacity of the Lung, ECG, Physical Examination, Orthostasis Test, Oxygen Saturation or Haemoccult Test
Description: Clinically relevant abnormalities for clinical laboratory evaluation, vital signs, lung function, carbon monoxide Diffusing Capacity Of the Lung (DLCO), Electrocardiogram (ECG), physical examination, orthostasis test, oxygen saturation or haemoccult test
Time Frame: From administration of study drug until end-of-study visit, up to 10 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Cmax
Description: Maximum measured concentration of the analyte in plasma (Cmax).
  The analysis population was the pharmacokinetic (PK) set which included all subjects randomised and treated with study medication who provided at least 1 evaluable observation for a PK endpoint of Area Under the Concentration-time Curve from 0 to infinity (AUC0-inf), Area Under the Concentration-time Curve from 0 to the last quantifiable data point (AUC0-tz) and Cmax and who had no important protocol violations relevant to the evaluation of PK.
Time Frame: Before drug administration and 15minutes (min), 30min, 45min, 1hour (h), 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 34h, 48h and 72h (for doses >=50mg only) after drug administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol/L | 1.36 (23.3) [0.50 to 1.00] | 1.66 (33.2) [0.50 to 1.00] | 2.83 (33.5) [0.25 to 4.00] | 7.33 (19.4) [0.75 to 4.00] | 23.5 (60.0) [0.50 to 4.00] | 52.6 (32.9) [0.25 to 4.00] | 202 (68.5) [0.25 to 6.00] | 459 (69.0) [0.50 to 2.00] | 984 (24.1) [0.75 to 1.52] | 1850 (16.4) [0.50 to 1.00]
Statistical Analysis 1: Comparison: BI 113608 0.5mg vs BI 113608 1mg vs BI 113608 2mg vs BI 113608 5mg vs BI 113608 10mg vs BI 113608 20mg vs BI 113608 50mg vs BI 113608 100mg vs BI 113608 150mg vs BI 113608 200mg; This was non confirmatory testing (Single dose). Dose proportionality of BI 113608 (powder in bottle (PIB)) for Cmax was analysed; Test type: Superiority or Other; Slope = 1.2472, 95% CI 2-sided [1.1831 to 1.3112], Standard Error of Mean 0.0320 — Dose proportionality was explored using the power model (ANCOVA). The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale. Standard Error of the mean is actually the Standard Error of the slope

3. Secondary Outcome: Tmax
Description: Time from dosing to maximum measured concentration of the analyte in plasma (Tmax)
Time Frame: as for outcome 2
Population: PK set
Measure: Median (Full Range); unit: Hours
Arm/Group | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 0.63 [0.50 to 1.00] | 0.88 [0.50 to 1.00] | 2.25 [0.25 to 4.00] | 1.75 [0.75 to 4.00] | 1.00 [0.50 to 4.00] | 1.10 [0.25 to 4.00] | 0.76 [0.25 to 6.00] | 0.63 [0.50 to 2.00] | 0.75 [0.75 to 1.52] | 0.63 [0.50 to 1.00]

4. Secondary Outcome: AUC0-tz
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz)
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol*h/L | 6.15 (23.7) [0.50 to 1.00] | 11.4 (62.3) [0.50 to 1.00] | 19.1 (30.7) [0.25 to 4.00] | 53.9 (18.3) [0.75 to 4.00] | 142 (24.2) [0.50 to 4.00] | 304 (24.7) [0.25 to 4.00] | 861 (34.8) [0.25 to 6.00] | 1990 (40.6) [0.50 to 2.00] | 4240 (18.2) [0.75 to 1.52] | 5950 (25.9) [0.50 to 1.00]
Statistical Analysis 1: Comparison: BI 113608 0.5mg vs BI 113608 1mg vs BI 113608 2mg vs BI 113608 5mg vs BI 113608 10mg vs BI 113608 20mg vs BI 113608 50mg vs BI 113608 100mg vs BI 113608 150mg vs BI 113608 200mg; This was non confirmatory testing (Single dose). Dose proportionality of BI 113608 (PIB) for AUC 0- tz was analysed; Test type: Superiority or Other; Slope = 1.1626, 95% CI 2-sided [1.1195 to 1.2057], Standard Error of Mean 0.0215 — Dose proportionality was explored using the power model (ANCOVA). The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale. Standard Error of the mean is actually Standard Error of the slope

5. Secondary Outcome: AUC0-infinity
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity)
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol*h/L | 6.54 (23.3) [0.50 to 1.00] | 12.2 (60.3) [0.50 to 1.00] | 19.9 (28.7) [0.25 to 4.00] | 55.2 (18.8) [0.75 to 4.00] | 144 (23.2) [0.50 to 4.00] | 307 (25.2) [0.25 to 4.00] | 862 (34.7) [0.25 to 6.00] | 1990 (40.6) [0.50 to 2.00] | 4250 (18.2) [0.75 to 1.52] | 5960 (25.9) [0.50 to 1.00]
Statistical Analysis 1: Comparison: BI 113608 0.5mg vs BI 113608 1mg vs BI 113608 2mg vs BI 113608 5mg vs BI 113608 10mg vs BI 113608 20mg vs BI 113608 50mg vs BI 113608 100mg vs BI 113608 150mg vs BI 113608 200mg; This was non confirmatory testing (Single dose).Dose proportionality of BI 113608 (PIB) for AUC0-inf was analysed; Test type: Superiority or Other; Slope = 1.1510, 95% CI 2-sided [1.1080 to 1.1941], Standard Error of Mean 0.0215 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: t1/2
Description: Terminal half-life of the analyte in plasma (t1/2)
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 4.66 (22.4) [0.50 to 1.00] | 8.10 (38.0) [0.50 to 1.00] | 8.56 (17.5) [0.25 to 4.00] | 8.08 (39.6) [0.75 to 4.00] | 10.3 (24.2) [0.50 to 4.00] | 9.51 (26.6) [0.25 to 4.00] | 11.2 (7.54) [0.25 to 6.00] | 12.8 (11.2) [0.50 to 2.00] | 12.5 (15.6) [0.75 to 1.52] | 11.8 (12.9) [0.50 to 1.00]

7. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentage of participants with drug-related adverse events
Time Frame: From administration of study drug until end-of-study visit, up to 10 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 50.0 | 0.0 | 33.3

8. Primary Outcome: Assessment of Tolerability by the Investigator
Description: Assessment of tolerability by the investigator assessed according to the categories good, satisfactory, not satisfactory, bad and not assessable.
Time Frame: End of study visit, up to day 10
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants
  Good | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100
  Satisfactory | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not satisfactory | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bad | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not assessable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From administration of study drug until end-of-study visit, up to 10 days
Arm/Group | Placebo | BI 113608 0.5mg | BI 113608 1mg | BI 113608 2mg | BI 113608 5mg | BI 113608 10mg | BI 113608 20mg | BI 113608 50mg | BI 113608 100mg | BI 113608 150mg | BI 113608 200mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/20 | 3/6 | 1/6 | 1/6 | 0/6 | 3/6 | 0/6 | 0/6 | 4/6 | 0/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | BI 113608 0.5mg (N=6) | BI 113608 1mg (N=6) | BI 113608 2mg (N=6) | BI 113608 5mg (N=6) | BI 113608 10mg (N=6) | BI 113608 20mg (N=6) | BI 113608 50mg (N=6) | BI 113608 100mg (N=6) | BI 113608 150mg (N=6) | BI 113608 200mg (N=6)
Retrograde amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | BI 113608 0.5mg (N=6) | BI 113608 1mg (N=6) | BI 113608 2mg (N=6) | BI 113608 5mg (N=6) | BI 113608 10mg (N=6) | BI 113608 20mg (N=6) | BI 113608 50mg (N=6) | BI 113608 100mg (N=6) | BI 113608 150mg (N=6) | BI 113608 200mg (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.